CLINICAL TRIAL: NCT05345028
Title: Positive Effects of a Lecithin-based Delivery Form of Boswellia Serrata Extract in Acute Diarrhea of Adult Subjects
Brief Title: Boswellia Serrata Extract in Acute Diarrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda di Servizi alla Persona di Pavia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4806/11012022
Record Dates: First submitted 2022-04-12; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Acute Diarrhea; Boswellia Serrata

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Boswellia Phytosome (Active Comparator)
  Interventions: Dietary Supplement: lecithin-based delivery form of Boswellia serrata
- Placebo (Placebo Comparator)
  Interventions: Combination Product: Placebo

INTERVENTIONS:
Dietary Supplement: lecithin-based delivery form of Boswellia serrata — 250 mg for 5 days
  Arms: Boswellia Phytosome
Combination Product: Placebo — 250 mg for 5 days
  Arms: Placebo

SUMMARY:
Acute diarrhea is a frequent problem worldwide, mostly due to gastrointestinal infections or food poisoning. Boswellia serrata could be active in the treatment of acute diarrhea due to its an-ti-inflammatory, antispasmodic and antimicrobial activity.

ELIGIBILITY:
Inclusion Criteria:

* presence of acute diarrhea of mild to moderate severity

Exclusion Criteria:

* patients with long term diarrhea
* iatrogenic diarrhea
* symptoms of functional gut disease or severe inter-current diseases
* severe diarrhea and dehydration requiring hospitalization and intravenous treatment
* subjects with high temperature (> 38.5° C)
* subjects treated by other anti-diarrheal and antibiotic drugs in the last 24 hours
* severely malnourished subjects
* pregnant women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2021-05-24 (Actual); Study Completion 2021-09-07 (Actual)

PRIMARY OUTCOMES:
Stoppage of diarrhea | From baseline to 5 days
  the occurrence of the first formed stool or a period of 12 hours without any liquid or soft stools

SECONDARY OUTCOMES:
Self-assessed symptoms | After 5 days
  daily number of stools within 5 days of treatment
Self-assessed symptoms | After 5 days
  percentage of subjects without diarrhea within 5 days of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda di Servizi alla Persona, Pavia, Italy

IPD SHARING:
Plan to Share IPD: Undecided